CLINICAL TRIAL: NCT05238688
Title: Evaluation of the Efficacy of Ipsilateral High Thoracic Ultrasound-guided Erector Spinae Plane Block in Preventing Post-thoracotomy Shoulder Pain in Thoracic Cancer Surgeries: A Prospective Randomized Controlled Study
Brief Title: Efficacy of Ipsilateral High Thoracic Ultrasound-guided Erector Spinae Plane Block in Thoracic Cancer Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Muhammad Mahmoud Sami Salahaldin Megahed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AP2109-30108
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Thoracotomy; Erector Spinae Plane Block; Thoracic Cancer; Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Tea; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic Epidural Analgesia (TEA) group (Experimental): Patients in this group will receive Thoracic Epidural analgesia.
  Interventions: Procedure: Thoracic Epidural Analgesia (TEA) group
- Thoracic Epidural Analgesia and Erector Spinae Plane Block (ESPB) group (Experimental): Patients in this group will receive Thoracic Epidural analgesia in addition to high thoracic ultrasound-guided erector spinae plane block (ESPB).
  Interventions: Procedure: Thoracic Epidural Analgesia and Erector Spinae Plane Block (ESPB) group

INTERVENTIONS:
Procedure: Thoracic Epidural Analgesia (TEA) group — Under full aseptic conditions while the patient is in setting position, skin infiltration will be done with 2 ml of 1% lidocaine an 18-G Tuohy needle with a 20-G catheter (Perifix, B.Braun, Germany) will be inserted through the T6-T7 interspace, and the epidural space located using the loss of resistance technique. The catheter then advanced approximately 3 cm cephalic. A test dose of 3 ml of 1% lidocaine containing epinephrine in a ratio of 1:200,000 administered to detect unintentional intrathecal . After negative response, 15 ml of 0.25% epidural bupivacine will be injected and the patient will be turned to the supine position.
  Arms: Thoracic Epidural Analgesia (TEA) group
Procedure: Thoracic Epidural Analgesia and Erector Spinae Plane Block (ESPB) group — Thoracic Epidural Analgesia will be done at first. Then, the ultrasound probe will be placed longitudinally 2-3 cm lateral to the T2 spinous process in the sagittal line. The T2 spinous process will be identified by counting down anatomically from the vertebral prominens (C7), and the T2 transverse process will be visualized by counting down from the first rib via real-time ultrasound guidance. The erector spinae muscle will be visualized above the T2 transverse process. The needle will be inserted in a caudal cranial direction using the in-plane technique. A dose of 5 mL normal saline will be injected into the inter-fascial area between the erector spinae muscle and the transverse process for the correction of the injection site (hydro-dissection). After hydro-dissection, 15 mL of 0.25% bupivacaine will be injected here, and the linear spread of the solution will be visualized in the inter-fascial plane.
  Arms: Thoracic Epidural Analgesia and Erector Spinae Plane Block (ESPB) group

SUMMARY:
To evaluate the effectiveness of ultrasound guided Erector Spinae Plane Block (ESPB) in controlling post thoracotomy ipsilateral shoulder pain.

DETAILED DESCRIPTION:
The aim of thoracotomy surgery is to explore the thoracic cavity and manage different pathologies including pulmonary, diaphragmatic, mediastinal, esophageal and vascular pathologies. It can be performed posterolaterally, anterolaterally or even anteriorly.

Post-thoracotomy Ipsilateral Shoulder Pain could undermine pain management in the post-thoracotomy patient.

Erector spinae plane block is a relatively novel block and was first described for chronic thoracic neuropathic pain in 2016. It is an inter-fascial plane block, but it may be classified as a paraspinal block due to its mechanism of action and injection site. It has been reported for a variety of indications, as in thoracic neuropathic pain and in postoperative analgesia after major open abdominal surgery. Erector spinae plane block has been successfully used to treat chronic shoulder pain, and the local anesthetic spread was reported to reach the level of C3 when it was performed at T2.

Ultrasound imaging made the practice of regional anesthesia easier in visualization and identification of usual and unusual position of nerves, blood vessels, needle during its passage through the tissues, as well as deposition and spread of local anesthetics in the desired plane and around the desired nerve.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status class I and II.
2. Age ≥ 18 and ≤ 60 Years.
3. Patients undergoing thoracic surgery e.g.: metastatectomy, lobectomy, pneumonectomy or pleuro-pneumonectomy.

Exclusion Criteria:

1. Patient refusal.
2. Local infection at the puncture site.
3. Coagulopathy with the international normalized ratio (INR) ≥ 1.6: hereditary (e.g. hemophilia, fibrinogen abnormalities and deficiency of factor II) - acquired (e.g. impaired liver functions with prothrombin concentration less than 60 %, vitamin K deficiency & therapeutic anticoagulants drugs).
4. Unstable cardiovascular disease.
5. History of psychiatric and cognitive disorders.
6. Patients allergic to medication used.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with ipsilateral shoulder pain. | one hour postoperatively
  Percentage of patients with ipsilateral shoulder pain with a Visual Analogue Scale (VAS) ≥ 3 where (0 = no pain and 10 = severe pain) in the first postoperative hour.

SECONDARY OUTCOMES:
Time to first rescue analgesia | 24 hours postoperatively
  Time to first analgesic request after surgery in the form of intravenous morphine in a dose (0.05 mg/kg)
Changes in postoperative heart rate | Preoperatively, intraoperatively, and 24 hours postoperatively
  Heart rate will be recorded before block performance and before induction of anesthesia, intraoperatively every 10 min till the end of surgery and after surgery at T (30 min in Post-Anesthesia Care Unit (PACU), 2, 4, 6, 12, 24 hours).
Changes in postoperative in mean arterial blood pressure | Preoperatively, intraoperatively, and 24 hours postoperatively.
  Mean arterial blood pressure will be recorded before block performance and before induction of anesthesia, intraoperatively every 10 min till the end of surgery and after surgery at T (30 min in Post-Anesthesia Care Unit (PACU), 2, 4, 6, 12, 24 hours).
Total intra-operative fentanyl consumption. | intraoperatively
  In case of an elevation of heart rate or mean arterial blood pressure ≥ 20% of the baseline will be treated by fentanyl 0.5 μg / kg.
Changes in postoperative oxygen saturation | 24 hours postoperatively
  Mean oxygen saturation at predetermined time intervals (1, 2, 6, 12 and 24 hours).
Complications occurrence | 24 hours postoperatively
  Adverse events as bradycardia, hypotension, failed block, local anesthetic toxicity, drowsiness and dizziness.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Megahed, MSc, Principal Investigator — Cairo University
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
This study will be available upon a reasonable request from the corresponding author.
Supporting Information: Study Protocol
Time Frame: One year after the end of the study.